CLINICAL TRIAL: NCT00116649
Title: Open-Label Safety and Pharmacokinetic Study of AldaraTM (Imiquimod) Cream, 5% for One, Two, or Three Treatment Cycles to Surface Areas Greater Than 25 cm2 With Actinic Keratosis
Brief Title: Open-Label Safety Study to Evaluate Imiquimod Cream, 5% for Large Areas of Actinic Keratosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Graceway Pharmaceuticals, LLC (Industry)
Responsible Party: Sharon Levy, MD VP Product Development, Graceway Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1520-IMIQ
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Results first posted 2008-11-25 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Keratosis
Keywords: actinic keratosis lesions large head torso extremities; actinic keratosis
MeSH Terms: conditions — Keratosis; Keratosis, Actinic | interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aldara 5% (Experimental): Aldara® (imiquimod) cream, 5% supplied in 250 mg single-use packets.
  Interventions: Drug: imiquimod cream

INTERVENTIONS:
Drug: imiquimod cream — imiquimod 5% cream applied in doses ranging from one packet (12.5 mg) to 6 packets (75 mg) to either single or multiple body regions for up to 3 cycles
  Other Names: Aldara® (imiquimod) cream 5%

SUMMARY:
Actinic keratosis (AK) is a skin condition that shows up on skin routinely exposed to the sun, such as the face, scalp, shoulders, chest, back, arms, and hands. The purpose of this study is to evaluate the safety of one, two, or three cycles of imiquimod for the treatment of AK. The AK lesions treated can be in adjacent and nonadjacent areas of the head, torso, and extremities. The total surface area for the AK lesions must be greater than 25 cm2. The secondary objective is to evaluate the effectiveness of treatment with imiquimod in people with large surface areas of AK.

DETAILED DESCRIPTION:
This was a Phase 4, open-label, single-arm, multicenter study in male and female subjects aged 18 years or older with clinically diagnosed AK lesions, conducted at 31 investigational sites in the United States.

This study assessed the safety of imiquimod as a treatment for AK applied in doses ranging from one packet 12.5 mg) to 6 packets (75 mg) to either single or multiple body regions for up to 3 cycles, depending upon treatment success and AK lesion recurrence. Eligible subjects applied imiquimod 5% cream prior to normal sleeping hours 2 days per week to at least 4 clinically typical, visible, discrete, nonhypertrophic AK lesions in contiguous or noncontiguous treatment areas totaling greater than 25 cm2 at baseline. Multiple treatment areas could be exposed (i.e., head, torso and/or extremities), with the number of packets determined by the investigator but not to exceed one packet for each 25 cm2 treatment area, up to a maximum of 6 packets per dose. In each treatment cycle, dosing was to continue for 16 weeks (approximately 4 months), as instructed by the investigator, followed by a 2-month, treatment-free follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years of age.
* Have greater than 25 cm2 total treatment area(s) containing at least 4 actinic keratosis lesions.

Exclusion Criteria:

* Have any skin condition in the treatment area that may be made worse by treatment with imiquimod (e.g., rosacea, psoriasis, atopic dermatitis, eczema).
* Have received specific treatments/medications in the treatment area(s) within the designated time period prior to study treatment initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2005-06; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Levy, MD, Study Director — Graceway Pharmaceuticals
Locations (30):
- United States (30):
  - Phoenix, Arizona
  - Encino, California
  - Los Angeles, California
  - Riverside, California
  - San Diego, California
  - Santa Monica, California
  - Denver, Colorado
  - New Britain, Connecticut
  - Coral Gables, Florida
  - Hollywood, Florida
  - Miami, Florida
  - West Palm Beach, Florida
  - Arlington Heights, Illinois
  - Indianapolis, Indiana
  - Metairie, Louisiana
  - Boston, Massachusetts
  - Chaska, Minnesota
  - Henderson, Nevada
  - Reno, Nevada
  - New York, New York
  - High Point, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Portland, Oregon
  - Flourtown, Pennsylvania
  - Arlington, Texas
  - San Antonio, Texas
  - Woodbridge, Virginia
  - Spokane, Washington
  - Milwaukee, Wisconsin

REFERENCES:
- [Result] Del Rosso JQ, Sofen H, Leshin B, Meng T, Kulp J, Levy S. Safety and Efficacy of Multiple 16-week Courses of Topical Imiquimod for the Treatment of Large Areas of Skin Involved with Actinic Keratoses. J Clin Aesthet Dermatol. 2009 Apr;2(4):20-8. PMID 20729935

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study start - 14 July 2005 at 31 study centers 500 subjects were planned, with up to 15 subjects enrolled at each study center; however, some study centers were unable to enroll 15 subjects, so active centers were asked to enroll additional subjects.
Pre-assignment Details: Open-label study - subjects were required to be at least 18 years of age and to have greater than 25 centimeters squared total treatment area(s) containing at least 4 clinically typical, visible, discrete, nonhypertrophic Actinic Keratosis lesions without any dermatological disease and/or condition in the treatment or surrounding area.
Groups:
- Aldara (Imiquimod) Cream: Aldara (imiquimod) Cream 5%
Period: Overall Study
Arm/Group | Aldara (Imiquimod) Cream
Started | 551 (586 screened (34 not eligible) 552 enrolled 551 study population (1 subject not treated))
Completed | 396
Not Completed | 155
Not completed — Adverse Event | 20
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 32
Not completed — Withdrawal by Subject | 68
Not completed — Local Skin Reaction | 9
Not completed — Various Reasons | 18
Not completed — Protocol Specified | 7

BASELINE CHARACTERISTICS:
Arm/Group | Aldara (Imiquimod) Cream
Number analyzed (Participants) | 551
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 207
  >=65 years | 344
Age Continuous [Mean (Standard Deviation); unit: years] | 67.5 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114
  Male | 437
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22
  Not Hispanic or Latino | 529
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 551
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 551
Baseline actinic keratosis lesion count [Mean (Standard Deviation); unit: actinic keratosis lesions] | 45.5 (2.36)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event
Description: Adverse events that occurred between the first day of exposure to the study cream and study discharge were summarized. Adverse events - any untoward medical occurrence in a subject that is temporally related to protocol procedures, including the administration of a pharmaceutical product at any dose, but which does not necessarily have a causal relationship with the treatment.
Time Frame: from first dose up to 18 months
Population: There were 551 subjects in the Safety population, which consisted of the enrolled subjects who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Aldara (Imiquimod) Cream
Number analyzed (Participants) | 551
participants | 472

2. Secondary Outcome: Percent Reduction From Baseline to the Final Follow-up in Total Actinic Keratosis Lesion Count
Description: Percent reduction = (total baseline AK lesion count - total final lesion count)x100/ total baseline AK lesion count
Time Frame: At Month 18
Population: The ITT population (n=526) consisted of the Safety population who had at least one scheduled primary efficacy assessment at a post-baseline visit
Measure: Mean (Standard Deviation); unit: percent reduction
Arm/Group | Aldara (Imiquimod) Cream
Number analyzed (Participants) | 526
percent reduction | 80.2 (1.55)

ADVERSE EVENTS:
Time Frame: Adverse events that occurred between the first day of exposure to the study cream up until study discharge were reported. Expsure could be up to three 16-week treatment cycles depending upon treatment success and AK lesion recurrence.
Description: Reporting of AEs by subjects was recorded. Local skin reactions (LSRs) in the treatment areas were also evaluated. These were erythema, edema, weeping/ exudate, vesicles, erosion/ulceration, flaking/scaling/dryness, and scabbing/crusting. Other skin-related reactions not listed, such as burning, itching, bleeding, etc., were documented as AEs.
Arm/Group | Aldara (Imiquimod) Cream
Serious Adverse Events (participants affected / at risk) | 39/551
Other Adverse Events (participants affected / at risk) | 472/551
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aldara (Imiquimod) Cream (N=551)
Bradycardia (Cardiac disorders) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myocardial infarction (Cardiac disorders) | 4 (4)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 4 (4)
Bacteraemia (Infections and infestations) | 1 (3)
Cardiac disorder (Cardiac disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Arteriosclerosis (Vascular disorders) | 2 (3)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Device failure (Injury, poisoning and procedural complications) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Intrervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Chest pain (General disorders) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Intervertebral disk protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aldara (Imiquimod) Cream (N=551)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 168 (168)
Application site pruritus (Skin and subcutaneous tissue disorders) | 127 (127)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 83 (83)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 82 (82)
Skin lesion (Skin and subcutaneous tissue disorders) | 59 (59)
Application site irritation (General disorders) | 48 (48)
Seborrhoeic Keratosis (Skin and subcutaneous tissue disorders) | 42 (42)
Fatigue (General disorders) | 34 (34)
Skin Papilloma (Skin and subcutaneous tissue disorders) | 33 (33)
Application site pain (General disorders) | 30 (30)
Upper respiratory tract infection (Infections and infestations) | 27 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No